CLINICAL TRIAL: NCT00257829
Title: Improving Tumor Oxygenation in Cervical Cancer With Methazolamide
Brief Title: Improving Tumor Oxygenation in Cervical Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was closed due to lack of funding.
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Chao Family Comprehensive Cancer Center, Cancer Center, University of California, Irvine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 03-41
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Methazolamide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Methazolamide
Drug: Cisplatin

SUMMARY:
The Phenomenon of Tumor Hypoxia Many solid tumors are relatively resistant to treatment with ionizing radiation and certain chemotherapeutic agents such as anthracyclines that are affected adversely by acidic pH. These effects have primarily been attributed to the presence of hypoxic cells within the tumor. The relevance of hypoxia with respect to failure of radiotherapy to cure certain malignancies has had a chequered history. However, in recent years the evidence that hypoxia plays a central role in relative radioresistance has become more compelling.

Since approximately two-thirds of all women suffering from cervical carcinoma receive radiation as a component of their therapy, an enhanced understanding of the interactions between hypoxia and radiation as a component of their therapy, an enhanced understanding of the interactions between hypoxia and radiation resistance is critical to improving outcome among those with cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* The subject will have a malignant tumor of the cervix which is not curable by surgery in which it has been determined the subject is to receive the standard care of treatment of radiation therapy and chemotherapy.
* The subject must have adequate bone marrow function, renal function, hepatic function and neurologic function.
* The subject should be free of active infection requiring antibiotics.
* The subject must have signed the approved informed consent
* If the subject is of childbearing age, they must have a negative urine pregnancy test with effective contraception
* The subject must have met pre-entry requirements

  1. Physical examination to include pelvic examination, blood counts, assessment of liver and kidney status through blood studies
  2. A serum pregnancy test
  3. Detectable tumor will be measured.

Exclusion Criteria:

* The subject has not been clinically staged for their cancer
* The subject has evidence of or is being treated for an active infection
* The subject cannot perform the appropriate follow-up or complete the study for whatever reason.
* The subject has not consented to an additional tumor biopsy and MRI after my seven days of treatment with methazolamide
* The subject has evidence of chronic obstructive pulmonary disease
* The subject is currently breastfeeding
* The subject is pregnant
* The subject takes aspirin chronically
* The subject has a history of Stevens-Johnson syndrome
* The subject has not signed the approved informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-07; Primary Completion 2006-09-20 (Actual); Study Completion 2006-09-20 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility in improving tumor oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Devansu Tewari, MD, Principal Investigator — Chao Family Comprehensive Cancer Center